CLINICAL TRIAL: NCT06340321
Title: Impact of Metabolic Flexibility on Changes in Metabolic Health
Acronym: METPROS
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Rodrigo Fernandez-Verdejo, Visiting Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-081
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Insight study cohort: The proposed study will include the individuals who participated in the baseline assessment of the InSight study at Pennington Biomedical in 2008-2009. These participants were not subjected to any intervention.
  Interventions: Diagnostic Test: Metabolic flexibility in the fasted state; Other: Metabolic flexibility in euglycemic-hyperinsulinemic clamp; Other: Metabolic flexibility in the metabolic chamber

INTERVENTIONS:
Diagnostic Test: Metabolic flexibility in the fasted state — Measured at baseline during the InSight study (2008-2009). Calculated as the respiratory exchange ratio in the fasting state adjusted for the circulating concentrations of free fatty acids
Other: Metabolic flexibility in euglycemic-hyperinsulinemic clamp — Measured at baseline during the InSight study (2008-2009). Calculated as the change in respiratory exchange ratio adjusted for glucose disposal rate
Other: Metabolic flexibility in the metabolic chamber — Measured at baseline during the InSight study (2008-2009). Calculated as the difference between awake respiratory exchange ratio (from 8 a.m. to 11 p.m.) and sleeping respiratory exchange ratio during a 23-hour stay in the metabolic chamber

SUMMARY:
Metabolic flexibility is the capacity to adapt fuel oxidation to fuel availability so that ATP synthesis can match its cellular demands. Thus, for example, increases in glucose availability after a meal would increase glucose oxidation, while increases in lipid availability during fasting would increase lipid oxidation. Enhanced metabolic flexibility has been proposed to protect humans from metabolic diseases. Nevertheless, most studies examining associations between metabolic flexibility and metabolic health outcomes have used cross-sectional designs. Whether impaired metabolic flexibility causes or results from metabolic health impairment is thus unclear.

In this study, the investigators will use the data from a study conducted approximately 16 years ago in healthy participants without obesity. Using the data already collected in that study, the metabolic flexibility of each participant will be calculated. To test the association between metabolic flexibility and the change in metabolic health, the investigators will call back all the participants for a single follow-up visit to reassess several metabolic health outcomes. Thus, the main aim of the study is to test the association between metabolic flexibility and the change in metabolic health outcomes after 16 years in humans.

DETAILED DESCRIPTION:
Metabolic flexibility is the capacity to adapt fuel oxidation to fuel availability so that ATP synthesis can match its cellular demands. Thus, for example, increases in glucose availability after a meal would increase glucose oxidation, while increases in lipid availability during fasting would increase lipid oxidation. Enhanced metabolic flexibility has been proposed to protect humans from ectopic lipid accumulation and the subsequent development of insulin resistance and metabolic syndrome.

In humans, metabolic flexibility is assessed by measuring relative macronutrient oxidation (i.e., lipids and carbohydrates) in response to metabolic challenges that increase glucose or lipid availability. The respiratory exchange ratio (RER = CO2 production / O2 consumption) is used to determine relative macronutrient oxidation. The euglycemic-hyperinsulinemic clamp is a widely used challenge to assess metabolic flexibility as it increases glucose availability and thus relative glucose oxidation. Recently, other methods have been proposed to assess metabolic flexibility, including the relative lipid oxidation during an overnight fast or the difference between 24-hour RER and sleeping RER in non-exercise, energy balance conditions while staying in a metabolic chamber. The method most relevant for assessing the influence of metabolic flexibility and its effects on metabolic health outcomes is unknown.

The influence of metabolic flexibility on metabolic health outcomes remains uncertain. The lack of agreement across studies is explained by the variability in the metabolic challenges, differences in the analytical approach to compute metabolic flexibility, and the loose use of the metabolic flexibility concept in the context of many different phenomena. Moreover, most studies examining associations between metabolic flexibility and metabolic health outcomes have used cross-sectional designs. Whether impaired metabolic flexibility causes or results from metabolic health impairment is thus unclear. Longitudinal studies using well-controlled methods are required to determine the impact of metabolic flexibility on prospective metabolic health.

In this pilot and feasibility study, the investigators will use the data from a study conducted 16 years ago in 88 healthy participants without obesity (InSight study at Pennington Biomedical). The study included an euglycemic-hyperinsulinemic clamp, an overnight fasting assessment, a 24-hour stay in a metabolic chamber, and the measurement of metabolic health outcomes. Using the data already collected in the InSight study, the metabolic flexibility of each participant in the euglycemic-hyperinsulinemic clamp, the overnight fast, and the metabolic chamber will be calculated. To test the association between metabolic flexibility(ies) and the change in metabolic health outcomes, the investigators will call back all the participants for a single follow-up visit to reassess the metabolic health outcomes including body mass index, body composition, blood pressure, HOMA-IR, and the circulating concentrations of glucose, triglycerides, and cholesterol. Such data will shed light on the most informative method to assess metabolic flexibility in relationship to specific metabolic health outcomes. The investigators will use these preliminary data to design and power future projects to be submitted for funding to scientific federal agencies.

Our specific aims are to:

1. Test the association between metabolic flexibility in response to a euglycemic-hyperinsulinemic clamp and the change in metabolic health outcomes after 16 years in humans.
2. Test the association between metabolic flexibility in response to overnight fasting and the change in metabolic health outcomes after 16 years in humans.
3. Test the association between metabolic flexibility in response to a 24-hour stay in a metabolic chamber and the change in metabolic health outcomes after 16 years in humans.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who participated in the InSight study at Pennington Biomedical in 2008-2009.

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding, have been pregnant in the last 12 months, and/or were breastfeeding in the last 6 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who participated in the InSight study at Pennington Biomedical in 2008-2009. Such study enrolled healthy men and women aged 20-36 years, with a body mass index <27.5 kg/m2, and a fasting glycemia <126 mg/dL.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Glucose | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Circulating concentration of glucose in mg/dL
Total cholesterol | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Circulating concentration of cholesterol in mg/dL
HDL cholesterol | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Circulating concentration of HDL cholesterol in mg/dL
LDL cholesterol | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Circulating concentration of LDL cholesterol in mg/dL
Triglycerides | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Circulating concentration of triglycerides in mg/dL
HOMA-IR | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Homeostatic Model of Assessment of Insulin Resistance computed from the circulating concentrations of glucose and insulin
Blood pressure | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Including systolic, diastolic, and mean blood pressure in mmHg
Waist circumference | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Measured in cm
Body mass index | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Calculated from the ratio between the weight and height, and expressed in kg/m2
Body fat percentage | At baseline (in 2008-2009) and after approximately 16 years (2024-2025)
  Measured by DXA and expressed as percentage of body weight

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fernández-Verdejo, PhD, Principal Investigator — Pennington Biomedical Research Center; Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center; Leanne Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected will be shared upon appropriate request as part of the NORC repository of Pennington Biomedical Research Center
Supporting Information: Study Protocol, ICF
Time Frame: After publication of the results for the main outcome
Access Criteria: Upon appropriate request
URL: https://my.pbrc.edu/NORC/NORCRepository/Landing/